CLINICAL TRIAL: NCT01308528
Title: A Non-Inferiority Study of Enoxaparin Cristalia in Relation With Enoxaparin Sanofi-Aventis for Prophylaxis Against Venous Thromboembolism in Patients With High-Risk to Develop Thromboembolic Disease Undergoing Geral Abdominal Surgery
Brief Title: Prophylactic Use of Sodium Enoxaparin for Venous Thromboembolism in High-Risk Abdominal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRT062
Record Dates: First submitted 2011-03-01; First posted 2011-03-04 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Venous Thromboembolism
Keywords: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — enoxaparin sodium; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium enoxaparin (Experimental): Endocris - 40 mg/0,4mL
  Interventions: Drug: Sodium enoxaparin
- sodium enoxaparin Clexane (Experimental): Clexane - 40 mg/ 0,4mL
  Interventions: Drug: Sodium Enoxaparin clexane

INTERVENTIONS:
Drug: Sodium enoxaparin — 40 mg/mL
  Other Names: Endocris
  Arms: Sodium enoxaparin
Drug: Sodium Enoxaparin clexane — clexane 40 mg/ 0,4 mL
  Other Names: clexane
  Arms: sodium enoxaparin Clexane

SUMMARY:
The purpose of this study is to compare the safety and security and efficacy of sodium enoxaparin Cristália Produtos Químicos Farmaceuticos Ltda - Endocris with Clexane (Sanofi-Aventis) to prevent Venous Thromboembolism in Patients With High-Risk to Develop Thromboembolic Disease Undergoing Geral Abdominal Surgery.

DETAILED DESCRIPTION:
This study is a requirement of Anvisa to add a new indication for off-label drug

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged above 18 years undergoing abdominal surgery with general high risk for developing venous thromboembolism;
* Who have provided their consent by signing the consent form.

Exclusion Criteria:

* Clinical evidence of Venous thromboembolism (VTE) in the selection;
* treatment requirement with anticoagulant Low Molecular Weight Heparin, Unfracted Heparin, oral anticoagulant
* suspicion or history of coagulumpathia
* Heparin, enoxaparin allergy or hypersensitiviy known to heparin, enoxaparin, but not restrict to thrombocytopenia and/or induce thombose by heparin ou enoxaparin (thrombocytopenia induce by heparin [TIH], thrombocytopenia associate with heparin [TAH] or thrombotic thrombocytopenia syndrome induce by heparin [STTIH]
* Active bleeding that can be increased by enoxaparin.
* Previous history of known intracranial hemorrhage
* Artery-venous malformation or a suspicion or known cerebral aneurism
* Spinal, Epidural ou lumbar puncture analgesia in the last 24 hours previous of the first dose of the administration of the enoxaparin.
* erosive diseases of the digestive tract especially gastroduodenal
* Uncontrolled hypertension (systolic blood pressure [BP]> 180mmHg or diastolic BP> 100 mm Hg) at randomization or clinical hypertensive urgency;
* bacterial endocarditis
* heart valve prosthesis
* characterized by severe renal insufficiency creatinine clearance <30 ml / min
* Intra-arterial thrombolic therapy
* Thrombolic therapy within 24 hours.
* Low Molecular Weight Heparin or Unfraction Heparin treatment with prophylactic dose over 48 hours before surgery or oral anticoagulant within 5 days before surgery
* disturbance of consciousness and coma
* Less than 6 months of expectative time life
* Chemical dependency
* Patient with anesthetic risk ASA III or ASA IV
* morbid obesity with Body Mass Index ≥ 40
* Chronic use of corticosteroids
* History of allergy to Unfraction Heparin, Low molecular weight heparin or pork products.
* History of severe allergic episode, systemic anaphylaxis, or major urticarial disease Steven-Johnson
* Participation in another clinical study within 12 months prior to inclusion
* Potentially fertile woman without β-HCG negative harvested until 48 hours before operation or not using acceptable contraception for participation in this study
* Changes the security checks up to 48 h before randomization:

  * Hemoglobin <10 mg / dL;
  * ALT or AST ≥ 2.5 times ULN;
  * Platelet count <100.000/mL;
  * INR ≥ 1.5;
* Any condition which in the opinion of the investigator, could lead to increased risk for the patient or who makes it inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of Sodium enoxaparin to demonstrate non-inferiority | 10 Days
  Evaluation of Prophylactic use of Sodium enoxaparin to demonstrate non-inferiority for Venous Thromboembolism in High-Risk Surgery in Abdominal

SECONDARY OUTCOMES:
Safety of sodium enoxaparine | 10 days
  comparision between Endocris (sodium enoxaparin - Cristalia Prod. Quim. Farm.) versus Clexane (sodium enoxaparine - Sanofi-Aventis) in High-Risk Abdominal Surgery.
Compare the incidence of venous thromboembolism and pulmonar embolism | 10 days
  Compare the incidence of venous thromboembolism and pulmonar embolism between 2 groups after 30 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gilson R de Araujo, PhD, Principal Investigator — Hospital Regional da Asa Norte
Locations (9):
- Brazil (9):
  - Hospital Regional da Asa Norte, Brasília, Federal District
  - Huning Instituto de Oftalmologia e Pesquisa HIOP/HRPC, Canoas, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundação de Desenvolvimento da Unicamp - FUNCAMP, Campinas, São Paulo
  - Hospital das Clínicas de Riberião Preto, Ribeirão Preto, São Paulo
  - Hospital Estadual Mario Covas, Santo André, São Paulo
  - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São Jósé Do Rio Preto, São Paulo